CLINICAL TRIAL: NCT05111470
Title: Analysis of the Kinematics of the Shoulder Complex in Sports "Overhead" Gestures Such as Kayaking Polo Throwing (Overhead)
Acronym: Overhead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A00494-53
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Kayak Polo; Overhead

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- kayak polo players (Experimental): Having a level of expertise greater than or equal to the national level 4
  Interventions: Other: Arm throws with his dominant arm

INTERVENTIONS:
Other: Arm throws with his dominant arm — Seated patient with different sensors on his naked torso. Patients will throw a ball with their dominant arm. The trajectories will be recorded by Vicon MX-40

SUMMARY:
The objective of this study is to analyze the throwing gesture specific to the kayak polo. A throw in a seated position with fixation of the pelvis (by the seat) and antepulsion of the hip ipsilateral to the throwing shoulder.

ELIGIBILITY:
Inclusion Criteria:

* free and informed consent signed
* Benefiting from a social protection insurance
* Over 18 years-old
* Male
* Having a level of expertise greater than or equal to the national level 4

Exclusion Criteria:

* Present during the study or have presented within the year any musculoskeletal pathology in the right and left shoulder.
* Have a body mass index greater than 30kg / m2 (to ensure sufficient accuracy to measure the movements of the scapula)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Glenohumeral and scapulothoracic angles | 1 hour
  Glenohumeral and scapulothoracic angles during throwing gestures with fixed pelvis associated with an initially antepulsed hip and free pelvis with the hip initially posteriorized

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France